CLINICAL TRIAL: NCT01693731
Title: Oral Health in Breast Cancer Survivors on Aromatase Inhibitors
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Linda Susan Taichman, Principal Investigator, University of Michigan
Other Study IDs: 5K23DEO21779; 5K23DE021779 (NIH); HUM00048451 (Other: UM MEDIRB)
Record Dates: First submitted 2012-09-18; First posted 2012-09-26 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Periodontal Disease; Quality of Life
Keywords: Breast cancer; Periodontal Diseases; Aromatase Inhibitors; Oral Health Related Quality of Life
MeSH Terms: conditions — Periodontal Diseases; Breast Neoplasms

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Each patient will have 5ml of blood collected at the visit. Saliva, and urine will also be collected at the study visit.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Aromatase Inhibitor: Postmenopausal women with breast cancer taking Arimidex, Aromasin, or Femara
- No Treatment: Healthy volunteer postmenopausal women not taking Aromatase Inhibitors

SUMMARY:
The purpose of this study is to determine how aromatase inhibitors (AIs) such as Arimidex, Aromasin or Femara affect a woman's oral health and oral health related quality of life. Patients, dental professionals and medical oncologists will benefit from a greater understanding of the best oral care follow up practices of breast cancer survivors using aromatase inhibitors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

This cross-sectional prevalence study seeks to investigate the incidence and severity of oral health changes, specifically of periodontal conditions, among breast cancer survivors and the ways in which these outcomes affect their quality of life.

Secondary

* To determine the prevalence and severity of oral conditions in postmenopausal women with early stage breast cancer using adjuvant AI therapy as compared to postmenopausal women not using adjuvant AI therapy.
* To determine if adjuvant AI therapy use is associated with greater alveolar bone loss or increased levels of bone turnover biomarkers in postmenopausal women with cancer undergoing adjuvant AI therapy compared to postmenopausal women not receiving AI therapy.
* To determine the oral health-related quality of life among postmenopausal women with early stage breast cancer who are receiving adjuvant AI therapy.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal as defined by NCCN (any of the following)

* Prior bilateral oophorectomy
* Age equal to or greater then 60 years of age
* Age less then 60 and amenorrheic for 12 or more months in the absence of chemotherapy, tamoxifen, toremifen or ovarian suppression and FSH and estradiol in the postmenopausal range
* If taking tamoxifen or toremifen and age less then 60y, then FSH and plasma estradiol level in postmenopausal ranges

Informed consent- Individuals capable of consenting and self administering the survey instrument Dentate- At least 15 teeth present.

AI users:

* Diagnosis of BCa- Histologic confirmed diagnosis of BCa: Stage 0, I, II, or III with no evidence of metastatic disease.
* Treatment- AI as clinically indicated (AI may be anastrozole, exemestane or letrozole) > 1 month. Subjects may have had prior tamoxifen or raloxifene. Subjects may have had chemotherapy and/or radiation therapy. Must be within the first year of consecutive AI therapy. If a subject started AI, discontinued, then restarted, they will be accepted into the study.

Controls:

* No Diagnosis of cancer.- Patients must not have a diagnosis of any cancer (Not including a history of localized thyroid or skin cancer).

Exclusion Criteria:

Medical history

* Metastatic BCa (AI treated group: fully resected locally recurrent disease is permitted if the patient has been rendered without evidence of disease).
* Significant psychiatric illness/social situations that would preclude completion of questionnaire.

Medications

* Chronic medications known to affect the periodontal status (calcium antagonist, anti-convulsives, immunosuppressives (> prednisone 7.5mg daily). NSAIDS and bisphosphonates are permitted.
* Premedication- Conditions that require antibiotic therapy will be evaluated on a case-by-case basis. (Patients taking prophylaxis for joint replacements will not be excluded.)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will have a sample of 300 postmenopausal women; 150 healthy women and 150 with early breast cancer using Aromatase Inhibitors
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Periodontal diseases | At the time of study visit

SECONDARY OUTCOMES:
Alveolar bone loss using salivary and serum-derived bone markers. | At the time of study visit
Oral Health Related Quality of Life (OHRQoL) assessed via questionnaire | At the time of study visit

CONTACTS AND LOCATIONS:
Overall Officials: L. Susan Taichman, RDH MPH PhD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Center For Oral Health Research (MCOHR), Ann Arbor, Michigan, United States